CLINICAL TRIAL: NCT06777160
Title: Predicting the Development of Bone Cement Implantation Syndrome in Arthroplasty Operations Using Artificial Intelligence Methods
Brief Title: Predicting Bone Cement Implantation Syndrome Using Artificial Intelligence Methods
Status: Recruiting | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Muhammed Cagatay Engin, associate professor doctor, Ataturk University
Other Study IDs: 499
Record Dates: First submitted 2025-01-05; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Bone Cement Implantation Syndrome
Keywords: CEMENT REACTION; ARTIFICIAL INTELLIGENCE; ARTHROPLASTY

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent arthroplasty and cement was used: For the operation of artificial intelligence modeling; First of all, the data to be entered into the system will be prepared. Some of the data will be entered manually (such as examination findings), some will be entered through the hospital information management system, and some will be converted into numerical form and entered manually (radiological reports). While data is being entered, critical criteria and panic values of each data will be introduced into the system. In this way, users will be warned when the system is activated.
  Interventions: Procedure: Collecting data from patients who underwent arthroplasty and cement was used

INTERVENTIONS:
Procedure: Collecting data from patients who underwent arthroplasty and cement was used — Collecting data that may change in cement reaction before, during and after surgery from patients who underwent arthroplasty and cement use and taught it to artificial intelligence.

SUMMARY:
This study aims to predict the development of bone cement syndrome, which may develop due to polymethylmethacrylate cement used to adhere the prosthesis to the bone in arthroplasty surgeries, which may cause intraoperative and postoperative mortality and morbidity, using artificial intelligence methods and to provide a sustainable life comfort to patients in the postoperative period with the standardization predicted in the long term.

DETAILED DESCRIPTION:
Since the prevalence of hip and knee osteoarthritis increases with age, orthopedic prosthesis operations are widely performed all over the world and in our country. In these surgeries, bone cement is used to ensure adhesion of the prosthesis to the bone. Bone cement implantation syndrome (BCIS) is a fatal complication of cemented bone surgery characterized by systemic hypotension, pulmonary hypertension, arrhythmias, loss of consciousness and cardiac arrest, most commonly occurring during cementing and prosthesis placement, and is increasingly being reported.

The syndrome is most commonly seen in cemented hemiarthroplasty after displaced femoral neck fractures, but also occurs in total hip and knee replacement surgery. Despite the publication of safety guidelines to reduce BCIS, it remains a common intraoperative complication with an overall incidence of up to 28% and is a major cause of intraoperative and postoperative morbidity and mortality.

The pathophysiology of BCIS is unclear, including hemodynamic instability as a result of changes in pulmonary and systemic vascular resistance, increased intramedullary pressure resulting in the incorporation of polymethyl methacrylate monomers into the circulation causing vasodilation, release of mediators from polymethyl methacrylate, release of fatty acids, and release of mediators from polymethyl methacrylate, Acute right ventricular failure, anaphylaxis, inflammatory and exothermic reaction, and complement activation may include one or a combination of acute right ventricular failure, anaphylaxis, inflammatory and exothermic reaction, and complement activation, which develops when cement and clot particles cause emboli in many organs in the body, especially in the pulmonary system, with increased pulmonary vascular resistance. Donaldson et al. developed a classification system for BCIS severity. Grade 0: no hypotension/hypoxia; Grade 1 moderate hypoxia (SpO2 < 94%) or hypotension [systolic blood pressure (SBP) > 20% decrease from baseline]; Grade 2 severe hypoxia (SpO2 < 88%) or hypotension (SBP > 40% decrease from baseline) or unexpected loss of consciousness; Grade 3 cardiovascular collapse requiring cardiopulmonary resuscitation.

Patients with BCIS grades 2 and 3 have been shown to have a 16-fold increase in 30-day postoperative mortality compared to those with BCIS grade 1. Most reports on BCIS focus on deaths and serious problems, and most cases of mild BCIS go unreported. Suspected BCIS should be treated with aggressive resuscitation and supportive care.

This risk may prompt some surgeons not to use cement in arthroplasty operations. Although cementless hemiarthroplasty eliminates this risk and saves an average operating time of 20 minutes, it is associated with serious complications. Patients undergoing uncemented hip arthroplasty implants are more likely to experience periprosthetic fractures as well as early revision. Uncemented arthroplasty has a 17-fold greater risk of periprosthetic fracture revision or aseptic revision due to loosening compared to cemented hip arthroplasty. Since additional surgery carries an additional risk of death, skipping the cementation step may also not be the best choice in these patients who are more likely to fall and undergo revision surgery.

Early detection of this complication and early intervention is crucial as it will reduce mortality. Prevention of BCIS includes identification of high-risk patients, preoperative optimization of patient risk factors and comorbidities, and good communication with the surgical team. In this way, the patient's comfort and life expectancy can be increased. The increasing number of patients needing and waiting for arthroplasty makes it difficult to identify high-risk patients, optimize patient risk factors and comorbidities preoperatively to prevent this potentially fatal complication.

The condition in which BCIS may occur is evaluated according to the results of analyzing the data obtained from retrospective and prospective data sets with complex biostatistical methods. In order to predict the complication, predictive factors associated with it are tried to be determined.

Spann et al. (2020) stated in their review study that machine learning can be used in analyzes beyond complex biostatistical methods. At this point, a decision support system created with artificial intelligence modeling will help in the early detection of this complication and thus serve as an important decision-support mechanism for clinicians by increasing the patient's comfort and life expectancy. However, it is not easy to assess at what level this complication will be predicted and reduced without implementing the system.

ELIGIBILITY:
Inclusion Criteria:

1. Total knee arthrplasties
2. Partial hip arthrplasty using cement
3. Total hip arthrplasty using cement
4. Patients ≥18 years old.

Exclusion Criteria:

Patients who do not want to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective study was conducted after obtaining the informed written consent of the patients and the ethics committee of Atatürk University Medical Faculty Research Hospital.
  on patients aged ≥18 years who underwent cemented total knee arthroplasty (TKA), cemented partial hip arthroplasty and cemented total hip arthroplasty It will be done.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-09-08 (Actual); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
collection of data-1 | 2 months
  General examination findings of the patient in the perioperative period, ASA score, whether the patient is female whether male or female, body mass index, age, whether mobility is decreased, whether assisted living, basic life parameters (operation blood pressure, pulse, respiratory rate, saturation, temperature, consciousness, orientation, etc.), the cause of the fracture (trauma, arthrosis, infection, necrosis, osteolysis, intertrochanteric fracture), type of surgery (total hip replacement, partial hip replacement, total knee replacement or revision surgery), medical history and medical history (cardiovascular disease, kidney disease, diabetes, stroke, peripheral vascular disease, arteriosclerosis, pulmonary hypertension, angina pectoris, congestive heart failure, COPD, cancer, dementia, arrhythmia, nicotine dependence, and the presence of previous myocardial infarction.
collection of data-2 | 2 months
  β-adrenergic blockers, diuretics, antiplatelet drugs, organic nitrates, calcium antagonists, ACE inhibitors, ARBs, acetylsalicylic acid, insulin, and warfarin and statin use), radiological evaluations (chest radiography), laboratory parameters (D-Dimer, IMA, IL-6, C-Peeptit, HbA1c, glucose, insulin, Ig E, NT Pro BNP, homocysteine, serotonin, adrenaline, noradrenaline, D vit, CK, CKMB, troponin, myoglobin, urea, uric acid, creatinine, AST, ALT, BIL, ALB, GGT, ALP, LDH, PT, PTT, INR, Sedim, CRP, fibrinogen, procalcitonin, TFT, HDL, LDL, TG, cholesterol, electrolytes and calcium, Mg, CA125, CA15-3, CA19
  -9, afp, CEA, hemogram, 5HT-2A receptor, GFR) and anaesthesia and surgery-related parameters (type of anaesthesia; general anaesthesia, local anesthesia) anaesthesia, volume of epidural anaesthetic used, type of local anaesthetic used, opioid use, duration of surgery, duration of anaesthesia, total blood loss
collection of data-3 | 2 months
  IMA measured at certain intervals after cementing. troponin-T measured at intervals, duration of hypotension, duration of hypoxia, medullary lavage, use of cement gun, vacuum cement Mixing and cementing pressure have been reported to be risk factors for the development of BCIS; these data will be collected throughout the study.
  When and which parameters will be performed will be determined by experienced physicians, and their results will be analysed according to their clinical experience.
  are interpreted by the algorithms they create.
artificial intelligence modeling | 1 months
  Artificial Intelligence model process steps The collected data will be made ready for artificial intelligence algorithms by going through the data preprocessing stage. In the feature extraction stage, simple feature extraction algorithms, kurtosis, skewness, local maximum, local minimum, hyperparameters, and principal component analysis processes will be applied. In the classification stage, a dataset is assigned to one of the predetermined classes that are different from each other. Classification algorithms learn which data to assign to which class from the given training set. Then it tries to assign the test data to the correct classes. Logistic regression, linear discriminant analysis, decision trees, Naive Bayes, the K-nearest neighbour algorithm, support vector machines, and random forest algorithms will be used in the classification phase. In the evaluation phase, the best model will be selected by creating an error matrix and interpreting the accuracy value of the model.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Faculty of Medicine, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is planned to share the data after it is collected and the artificial intelligence app is created.